NCT #: NCT03992131

# STATISTICAL ANALYSIS PLAN

SEASTAR: A Phase 1b/2, Open-label, Parallel Arm Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral Rucaparib in Combination with Other Anticancer Agents in Patients with a Solid Tumor

Arm A: rucaparib and lucitanib

PROTOCOL NUMBER: CO-338-098

VERSION: 1.0

**DATE FINAL:** 10 September 2021

**SPONSOR:** Clovis Oncology, Inc.

### **CONFIDENTIAL**

The information contained in this document is regarded as confidential and, except to the extent necessary to obtain informed consent, may not be disclosed to another party unless such disclosure is required by law or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# Approval Page




# TABLE OF CONTENTS

| TA | BLE O | F CONTENTS | 3 |
|----|---------|-----------------------------------------------|-----|
| LI | ST OF 1 | N-TEXT TABLES | 4 |
| LI | ST OF | APPENDICES | 4 |
| AF | BREV | IATIONS AND SPECIALIST TERMS | 5 |
| 1 | INT | RODUCTION | 7 |
| 2 | OV | ERALL STUDY DESIGN, OBJECTIVES, AND ENDPOINTS | 7 |
| | 2.1 | Study Design | 7 |
| | 2.2 | Study Objectives and Endpoints | 8 |
| | 2.3 Sa | mple Size Justification | 9 |
| 3 | GE | NERAL ANALYSIS CONVENTIONS | 9 |
| | 3.1 | Analysis Populations | 9 |
| 4 | PA | FIENT DISPOSITION | 9 |
| 5 | PRO | OTOCOL DEVIATIONS | 10 |
| 6 | DE | MOGRAPHICS AND BASELINE CHARACTERISTICS | |
| | 6.1 | Demographics | |
| | 6.2 | Baseline Clinical Characteristics | |
| | 6.3 | Medical History | |
| 7 | | SE-LIMITING TOXICITIES | |
| 8 | | STUDY DRUG EXPOSURE AND COMPLIANCE | |
| 9 | | OR AND CONCOMITANT MEDICATIONS | |
| 10 | | FICACY ANALYSIS | |
| 11 | | PLORATORY ANALYSIS | |
| 12 | | ARMACOKINETIC ANALYSIS | |
| 13 | | FETY ANALYSIS | |
| | 13.1 | Adverse Events | |
| | 13.2 | Clinical Laboratory Evaluations | |
| | | Vital Signs | |
| 14 | | ATISTICAL / ANALYTICAL ISSUES | |
| | 14.1 | Handling of Dropouts or Missing Data | |
| | 14.2 | Pooling of Centers in Multi-Center Studies | |
| | 14.3 | Multiple Comparison / Multiplicity | |
| | 14.4 | Examination of Subgroups. | |
| | 14.5 | Interim Analyses and Data Monitoring | |
| 15 | | FERENCES | |
| 16 | A D | DENDICES | 1.4 |

| I | JST | OF | In-t | EXT | TA | RI | ES |
|---|-----------|------------|------|-----|----|----|----|
| | / I L J I | <b>\</b> / | | | | | |

# LIST OF APPENDICES


Clovis Oncology 10 September 2021

## ABBREVIATIONS AND SPECIALIST TERMS

AE(s) adverse event(s)

ALT alanine aminotransferase
ANC absolute neutrophil count
AST aspartate aminotransferase

AUC<sub>0-last</sub> last quantifiable concentration

BID twice daily

CL/F plasma clearance

C<sub>max</sub> maximum observed concentration

C<sub>min</sub> minimum concentration

CR complete response

CRM cohort review meeting
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

ctDNA circulating cell-free tumor DNA

DBP diastolic blood pressure
DLT dose limiting toxicity
DOR duration of response

ECOG Eastern Cooperative Oncology Group

MTD maximum tolerated dose
NCI National Cancer Institute

ORR objective response per RECIST

PD progressive disease
PK pharmacokinetic(s)
PR partial response

QD once daily

RECIST Response Evaluation Criteria in Solid Tumors

RP2D Recommended Phase 2 dose

SAP statistical analysis plan SBP Systolic blood pressure

SD stable disease

SI International System of Units

StD standard deviation


Rucaparib CO-338-098A Statistical Analysis Plan Clovis Oncology 10 September 2021

TEAE treatment-emergent adverse event

 $T_{max}$  time to maximum concentration

ULN upper limit of normal


## 1 Introduction

This SAP describes the data summaries and any statistical analyses to be performed to assess the safety, efficacy, and pharmacokinetics (PK) of rucaparib (CO-338) for Clovis Oncology, Inc sponsored clinical study CO-338-098, entitled "SEASTAR: A Phase 1b/2, Open-label, Parallel Arm Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral Rucaparib in Combination with Other Anticancer Agents in Patients with a Solid Tumor."

This SAP addresses only the Phase 1b portion of Arm A of the study. The study reached the maximum rucaparib dose of 600 mg BID and a lucitanib dose of 6 mg QD. While the maximum tolerated dose (MTD) was not defined, the study was closed to further enrollment. The study will not continue to Phase 2 due to a change in priorities and no further clinical development of the lucitanib plus rucaparib combination is planned at this time. The analysis plan is therefore reduced from what was indicated in the protocol in order to support a abbreviated CSR. Results for Arm B of the Ph 1b part of the study are analyzed under a different SAP.

# 2 OVERALL STUDY DESIGN, OBJECTIVES, AND ENDPOINTS

### 2.1 STUDY DESIGN

For the Phase 1b portion of Arm A, the plan estimated 6 to 12 dose-escalation cohorts, with a minimum of 3 patients enrolled in each cohort, followed by an expanded evaluation of the recommended phase 2 dose (RP2D) in up to 10 additional patients. Dose escalation was to follow a 3+3 design.

The initial combination dose consisted of oral rucaparib 300 mg BID and oral lucitanib 4 mg QD, both administered continuously. In the initial program, the dose of rucaparib was to be escalated in 100 mg BID increments up to a maximum of 600 mg BID. A later protocol amendment allowed the final rucaparib dose to escalate from 400 to 600 mg BID. The dose of lucitanib was to be escalated in increments of 2 mg, up to a maximum dose of 10 mg QD.


### 2.2 STUDY OBJECTIVES AND ENDPOINTS

Because this study was terminated early, not all endpoints from the protocol will be analyzed. Table 1 outlines the objectives and endpoints planned per protocol for Phase 1b of Arm A. The final column includes the analyses to be included in the CSR.

Table 1. Primary, Secondary, and Exploratory Objectives and Endpoints for Phase 1b

| Primary Objectives | Primary Endpoints | Included in CSR |
|---|---|---|
| To evaluate the safety and tolerability of rucaparib in combination with lucitanib and to determine the MTD and/or the RP2D of the combination. | Incidence of AEs, clinical laboratory abnormalities, dose modifications, and blood pressure | Yes: AEs, some clinical laboratories, and dose modifications will be included |
| Secondary Objectives | Secondary Endpoints | |
| To characterize the PK of rucaparib and lucitanib when agents are co-administered. | Area under the curve from time zero to the last quantifiable concentration (AUC <sub>0-last</sub> ), maximum observed concentration (C <sub>max</sub> ), time to maximum concentration (T <sub>max</sub> ), and apparent plasma clearance (CL/F) | Not included in CSR |
| To evaluate the preliminary efficacy of rucaparib in combination with lucitanib in various solid tumors. | Objective response per RECIST v1.1 (ORR) | Yes |
| <b>Exploratory Objectives</b> | Exploratory Endpoints | |
| To assess tumor tissue biomarkers that correlate with response to the combination. | Not defined in protocol | Not included in CSR |
| To evaluate circulating cell-free tumor DNA (ctDNA) as a molecular marker of response to the combination. | Not defined in protocol | Not included in CSR |
| To evaluate biomarkers associated with resistance to the combination. | Not defined in protocol | Not included in CSR |
| To assess genomic changes over time in plasma and tumor samples. | Not defined in protocol | Not included in CSR |
| To determine steady-state exposure of rucaparib and lucitanib by sparse PK sampling. | Plasma concentration at trough (C <sub>min</sub> ) | Yes |


### 2.3 SAMPLE SIZE JUSTIFICATION

For Arm A Phase 1b, it was estimated that up to 55 patients would be enrolled following a standard 3+3 design, dependent upon the occurrence of safety findings, specifically dose limiting toxicities (DLTs), observed at the different dose levels. Nineteen subjects were enrolled before the study was terminated.

## 3 GENERAL ANALYSIS CONVENTIONS

Quantitative variables will typically be summarized using frequencies and percentages for appropriate categorizations and may also be summarized using descriptive statistics. For variables summarized with descriptive statistics, the following will be presented: N, mean, standard deviation (StD), median, minimum, and maximum. Categorical variables will be presented using frequencies and percentages.

Baseline is defined as the last measurement on or prior to the first dose of rucaparib administration, unless otherwise specified.

All statistical analyses will be conducted with the SAS® System, Version 9.4 or higher.

### 3.1 ANALYSIS POPULATIONS

The following analysis populations are defined for the study:

**Safety Population**: All patients who have received at least 1 dose of rucaparib or lucitanib.

**DLT-evaluable Population**: All patients in Phase 1b who have either received at least 80% of the planned doses of rucaparib and lucitanib without having experienced a DLT or who experienced a DLT during Cycle 1. If a patient withdrew from the study without having met any of these criteria, then an additional patient was enrolled in that dose cohort.

**Efficacy Population**: All patients who have received at least 1 dose of rucaparib or lucitanib and who have measurable disease per RECIST v1.1 at baseline.

**PK-Evaluable Population**: all patients who have received at least one dose of rucaparib or lucitanib and have had at least one measurable concentration.

# **4 PATIENT DISPOSITION**

Patient disposition will be summarized using frequency counts and the corresponding percentages. The number of patients in each analysis population, number of patients discontinued, and the primary reason for treatment discontinuation will be summarized.


## 5 PROTOCOL DEVIATIONS

The number of patients with major protocol deviations (eg, inclusion or exclusion criteria) will be determined prior to data base lock and will be summarized with frequencies and percentages or provided in a patient listing.

Protocol deviations will not be used to exclude any patients from the efficacy analyses.

### 6 DEMOGRAPHICS AND BASELINE CHARACTERISTICS

All demographics will be summarized for the safety population.

### 6.1 DEMOGRAPHICS

The demographic variables will be summarized with frequency tabulations and descriptive statistics. The demographic variables presented will include age, height, weight and sex using the following categorizations:

- Age (years):  $\leq 50$ , 51-60, 61-70, 71-80, 81-90,  $\geq 90$ ;
- Height (cm):  $\leq 75$ , > 75-100, > 100-125, > 125-150, > 150-175, > 175;
- Weight (kg):  $\leq 50$ , > 50-75, > 75-100, > 100-125, > 125-150, > 150
- Sex: Male, Female
- Race: American Indian or Alaskan Native, Asian, Black or African American, Native Hawaiian or Pacific Islander, White
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino
- Baseline ECOG: 0,1

### **6.2** Baseline Clinical Characteristics

HRD status will be listed.

### **6.3** MEDICAL HISTORY

Medical history events will not be analyzed.

## 7 DOSE-LIMITING TOXICITIES

A summary of the number of DLTs by dose level and a patient listing of all DLTs will be provided for the patients in the DLT-evaluable population. A DLT for Arm A is defined at any of the following events occurring in Cycle 1, according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0:


- Grade 3 or greater febrile neutropenia (i.e., fever > 38.3°C with Absolute Neutrophil Count (ANC) <  $1.0 \times 10^9$ /L) of any duration;
- Grade 3 thrombocytopenia (platelets  $< 50 \times 10^9/L$ ) with significant bleeding or Grade 4 thrombocytopenia (platelets  $< 25 \times 10^9/L$ )  $\ge 5$  days duration;
- Grade 4 anemia (i.e., life-threatening consequences; urgent intervention indicated) or any anemia (regardless of grade or severity) requiring a blood transfusion;
- Hypertension, defined as systolic blood pressure [SBP] ≥ 160 mmHg and/or diastolic blood pressure [DBP] ≥ 100 mmHg, that does not resolve to ≤ Grade 2 within 14 days despite optimized antihypertensive therapy, or any Grade 4 hypertension (hypertension with life-threatening consequences);
- Any nonhematological  $AE \ge Grade 3$ , with the exception of:
  - Nausea, vomiting, and diarrhea if well controlled by systemic medication and with duration < 48 hrs;
  - o Fatigue;
  - o Hyponatremia;
  - Grade 3 alanine aminotransferase (ALT) or aspartate aminotransferase (AST) not accompanied by a concomitant increase in total bilirubin above the upper limit of normal (ULN). Note: any Grade 4 ALT/AST is a DLT.

## 8 STUDY DRUG EXPOSURE AND COMPLIANCE

The following variables will be summarized:

- Duration of treatment (days)
- Duration of treatment (months)
- Number of cycles started
- Number of dose reductions
- Number of treatment interruptions
- Dose intensity

Duration of treatment will be calculated as 1+ the number of days from earliest study drug start date to date of last study drug discontinuation. Dose intensity will be calculated as the actual dose received divided by the assigned dose amount. Descriptive statistics and frequencies/percentages for appropriate categorizations will be used to summarize study drug exposure variables.

## 9 PRIOR AND CONCOMITANT MEDICATIONS

Prior and concomitant medications will not be analyzed in the CSR.

## 10 EFFICACY ANALYSIS

Efficacy analyses will be performed using the efficacy population.


Overall objective response to treatment according to RECIST v1.1 as assessed by the investigator will be listed along with target lesion measurements and response, non-target lesion response, and assessment of new lesions. Confirmation of a complete response (CR) or partial response (PR) is a response that is maintained and documented on a subsequent tumor assessment no less than 4 weeks after initial response. Duration of response (DOR) will also be calculated as the time from the date that a confirmed PR or CR is first recorded until the first date that progressive disease (PD) is documented per RECIST v1.1. Duration of stable disease (SD) will be calculated from the start of treatment to the first PD if the subject had a best response of SD.

A listing of all tumor scan details collected in the clinical database, including assessment of objective response and DOR will be provided.

## 11 EXPLORATORY ANALYSIS

Only the PK exploratory endpoint will be analyzed in the CSR. In all patients with at least one PK sample collected, the trough plasma rucaparib and lucitanib PK data ( $C_{min}$ ), summary statistics of  $C_{min}$  (N, mean, SD, minimum, median, max, CV%), and the mean ( $\pm$ SD) concentration versus time plot will be reported.

## 12 PHARMACOKINETIC ANALYSIS

The secondary PK analytical plan and analyses will be included in a separate PK report.

## 13 SAFETY ANALYSIS

The safety analyses will be performed using the safety population.

### 13.1 ADVERSE EVENTS

AEs will be classified using the MedDRA v. 24.0 classification system. The severity of the toxicities will be graded according to the National Cancer Institute (NCI) CTCAE v5.0 whenever possible. TEAEs are defined as AEs with onset date on or after the date of first dose of study medication until the date of the last study medication dose plus 28 days. Adverse events will be considered treatment-emergent if all or part of the date of onset of the AE is missing and it cannot be determined if the AE meets the definition for treatment-emergent.

The number and percentage of patients who experienced TEAEs for each system organ class and preferred term will be presented. Multiple instances of the TEAE in each system organ class and multiple occurrences of the same preferred term are counted only once per patient. The number and percentage of patients with at least one TEAE will also be summarized.

The incidence of TEAEs will also be summarized by relationship to study drug according to the following categories: "treatment-related," or "not treatment-related" for each study drug.


If a patient experiences multiple occurrences of the same AE with different relationship categories, the patient will be counted once, as a relationship category of treatment-related.

If a patient experiences multiple occurrences of the same AE with different toxicity grades, the patient will be counted once for the maximum (most severe) toxicity grade. AEs with a missing toxicity grade will be presented in the summary table with a toxicity grade of "Missing." For each toxicity grade, the number and percentage of patients with at least one TEAE of the given grade will be summarized.

Separate tables will be presented including but not limited to:

- All TEAEs;
- TEAEs by CTCAE grade;
- Grade 3 or greater TEAEs;
- Treatment-related TEAEs will be included in the following three categories of relatedness: related to rucaparib, related to lucitanib and related to either study drug. Relatedness will be analyzed, overall and by categories: CTCAE grade, grade 3 or greater, serious TEAEs, resulting in dose reduction, resulting in dose interruption, resulting in dose discontinuation, outcome of death;
- Serious TEAEs;
- TEAEs with an outcome of death;
- TEAEs leading to discontinuation of rucaparib only, lucitanib only, or either study drug;
- TEAEs resulting in interruption of rucaparib only, lucitanib only, or either study drug; and
- TEAEs resulting in reduction, delay, or interruption of rucaparib only, lucitanib only, or either study drug.

### 13.2 CLINICAL LABORATORY EVALUATIONS

Clinical laboratory evaluations include the continuous variables for hematology, chemistry, and urinalysis. The laboratory values will generally be presented in International System (SI) units. The on-treatment period will be defined as the time from earliest first dose to 28 days after the last dose of rucaparib or lucitanib, whichever is last. Hematology, chemistry and urinalysis values collected will be listed. Descriptive summaries, and all chemistry and urinalysis parameters, mentioned in the protocol will not be included in the analysis.

### 13.3 VITAL SIGNS

The on-treatment period will be defined as the time from first dose to 28 days after the last dose of study drug. Blood pressure measurements (systolic and dystolic) collected during the on-treatment period will be included in the summary tables. The blood pressure measurements collected after the on-treatment period will only be presented in the data listings.


The summary of blood pressure data will include descriptive statistics (N, mean, StD, minimum, median, and maximum) of the maximum, minimum, and last value during the ontreatment period. Summaries using descriptive statistics (N, mean, StD, minimum, median, and maximum) of the change from baseline to the maximum, minimum, and last value during the on-treatment period will also be given. The data will be presented separately for each treatment group and overall.

## 14 STATISTICAL / ANALYTICAL ISSUES

### 14.1 HANDLING OF DROPOUTS OR MISSING DATA

All data will be used to their maximum possible extent, but without any imputations for missing data.

### 14.2 POOLING OF CENTERS IN MULTI-CENTER STUDIES

All centers will be pooled for analysis.

### 14.3 MULTIPLE COMPARISON / MULTIPLICITY

No statistical comparisons will be performed.

### 14.4 EXAMINATION OF SUBGROUPS

Analyses of primary and secondary endpoints may be analyzed by starting dose. No additional subgroup analyses will be performed.

### 14.5 INTERIM ANALYSES AND DATA MONITORING

No formal interim analyses occurred outside standard Cohort Review Meetings (CRM). CRMs were held for the first 4 dose cohorts.

### 14.6 Analysis Included on CT.gov

Because enrollment was halted early with less than 20 subjects enrolled, only the primary endpoint will be included in CT.gov analyses


Clovis Oncology 10 September 2021

# 15 REFERENCES

1. Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45(2):228-47.


## 16 APPENDICES

### Appendix 1 Response Evaluation Criteria in Solid Tumors

The RECIST guidelines (Version 1.1) are described in Eisenhauer (2009)<sup>1</sup> and at http://www.eortc.be/Recist/Default.htm. A short summary is given below.

#### **Measurable Disease:**

<u>Tumor lesions</u>: measurable lesions are defined as those that can be accurately measured in at least 1 dimension (longest diameter to be recorded) with the following:

- A minimum size of 10 mm by CT scan (CT scan thickness no greater than 5 mm).
- A minimum size of 10 mm caliper measurement by clinical exam (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable).
- A minimum size of 20 mm by chest X-ray.

All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

Malignant lymph nodes: to be considered pathologically enlarged and measurable, a lymph node must be  $\geq 15$  mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be not greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

### Nonmeasurable Disease:

All other lesions (or sites of disease), including small lesions (longest diameter < 10 mm or pathological lymph nodes with  $\geq$  10 to < 15 mm short axis), as well as truly nonmeasurable lesions, are considered nonmeasurable disease. Lesions considered truly nonmeasurable include leptomeningeal disease, ascites, pleural/pericardial effusions, inflammatory breast disease, lymphangitic involvement of skin and lung, and abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.

#### **Bone Lesions**

Bone lesions, cystic lesion, and lesions previously treated with local therapy require particular comment. Bone scan, PET scan, or plain films are not considered adequate imaging techniques to measure bone lesions. However, these techniques can be used to confirm the presence or disappearance of bone lesions.

Lytic bone lesions or mixed lytic—blastic lesions with identifiable soft tissue components that can be evaluated by cross-sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the soft tissue component meets the definition of measurability described above.


Clovis Oncology 10 September 2021

Blastic bone lesions are nonmeasurable.

### **Cystic Lesions**

Lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor nonmeasurable) because they are, by definition, simple cysts.

Cystic lesions thought to represent cystic metastases can be considered as measurable lesions if they meet the definition of measurability described above. However, if noncystic lesions are present in the same patient, these are preferred as target lesions.

### **Lesions with Prior Local Treatment**

Tumor lesions situated in a previous irradiated area or in an area subjected to other locoregional therapy are usually not considered measurable unless there has been demonstrated progression in the lesion.

### **Target Lesions**

All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as target lesions and recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference by which to characterize the objective tumor response.

### **Nontarget Lesions**

RECIST criteria require unequivocal quantification of the changes in tumor size for adequate interpretation of the sum of target lesions. Consequently, when the boundaries of the primary are difficult to delineate, this tumor should not be considered a target lesion.

#### **Guidelines for Evaluation of Measurable Disease**

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination when both methods have been used to assess the antitumor effect of a treatment.


| Evaluation of Target L | Evaluation of Target Lesions |
|---|---|
| Complete Response | Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm. |
| Partial Response | At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. |
| Stable Disease | Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. |
| Progressive Disease | At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. |

Abbreviations: LD = longest diameter; PD = progressive disease.

| <b>Evaluation of Nontarget Lesions</b> | |
|---|---|
| Complete Response | Disappearance of all nontarget lesions and normalization of tumor marker level. |
| Stable Disease/Incomplete<br>Response | Persistence of 1 or more nontarget lesion(s) or/and maintenance of tumor marker level above the normal limits. |
| Progressive Disease | Appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions. |

If tumor markers are initially above the institutional ULN, they must normalize for a patient to be considered a complete responder.

### **Evaluation of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

| Evaluation of Best Overall Response | | | |
|---|---|---|---|
| Target Lesions | Nontarget Lesions | New Lesions | Overall Response |
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |


| <b>Evaluation of Best Overall Response</b> | | | | | |
|---|---|---|---|---|---|
| Targ | et L | esions | Nontarget Lesions | New Lesions | Overall Response |
| CR | | | Not evaluated | No | PR |
| PR | | | Non-PD or not evaluated | No | PR |
| SD | | | Non-PD or not evaluated | No | SD |
| Not Evaluated | | | Non-PD | No | NE |
| PD | | | Any | Yes or No | PD |
| Any | | | PD | Yes or No | PD |
| Any | | | Any | Yes | PD |
| CR | = | complete response | | | |
| NE | = | not evaluable. | | | |
| PD | = | progressive disease | | | |
| PR | = | partial response | | | |
| SD | = | stable disease | | | |

Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be classified as having symptomatic deterioration. Every effort should be made to document the objective progression, even after discontinuation of treatment.

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When the evaluation of CR depends on this determination, it is recommended that the residual lesion be investigated (fine needle aspiration/biopsy) prior to confirming the complete response status.

### **Confirmatory Measurement/Duration of Response**

### Confirmation

If a complete response (CR) or partial response (PR) is noted, confirmatory scans should be performed at least 4 weeks after response was first documented.

### **Duration of Overall Response**

The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or PD is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started).

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.


Rucaparib CO-338-098A Statistical Analysis Plan Clovis Oncology 10 September 2021

## **Duration of Stable Disease**

Stable disease (SD) is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.


NCT #: NCT03992131

# STATISTICAL ANALYSIS PLAN

SEASTAR: A Phase 1b/2, Open-label, Parallel Arm Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral Rucaparib in Combination with Other Anticancer Agents in Patients with a Solid Tumor

Arm B: rucaparib and IMMU-132 (sacituzumab govitecan)

PROTOCOL NUMBER: CO-338-098

VERSION: 1.0

**DATE FINAL:** 01 March 2021

**SPONSOR:** Clovis Oncology, Inc.

### **CONFIDENTIAL**

The information contained in this document is regarded as confidential and, except to the extent necessary to obtain informed consent, may not be disclosed to another party unless such disclosure is required by law or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# Approval Page




# TABLE OF CONTENTS

| | | F CONTENTS | |
|-----|------|-----------------------------------------------|-----|
| | | N-TEXT TABLES | |
| | | APPENDICES | |
| ABl | | ATIONS AND SPECIALIST TERMS | |
| 1 | | RODUCTION | |
| 2 | | ERALL STUDY DESIGN, OBJECTIVES, AND ENDPOINTS | |
| | 2.1 | Study Design | |
| | 2.2 | Study Objectives and Endpoints | |
| | | nple Size Justification | |
| 3 | | NERAL ANALYSIS CONVENTIONS | |
| | 3.1 | Analysis Populations | 8 |
| 4 | | TIENT DISPOSITION | |
| 5 | | OTOCOL DEVIATIONS | |
| 6 | | MOGRAPHICS AND BASELINE CHARACTERISTICS | |
| | 6.1 | Demographics | 9 |
| | 6.2 | Baseline Clinical Characteristics | 9 |
| | 6.3 | Medical History | 9 |
| 7 | | SE-LIMITING TOXICITIES | |
| 8 | STU | STUDY DRUG EXPOSURE AND COMPLIANCE 10 | |
| 9 | PRI | OR AND CONCOMITANT MEDICATIONS | 1( |
| 10 | EFF | ICACY ANALYSIS | 10 |
| 11 | EXF | PLORATORY ANALYSIS | 11 |
| 12 | PHA | ARMACOKINETIC ANALYSIS | 11 |
| 13 | SAF | ETY ANALYSIS | 11 |
| | 13.1 | Adverse Events | 11 |
| | 13.2 | Clinical Laboratory Evaluations | 12 |
| | 13.3 | Vital Signs | 12 |
| 14 | STA | TISTICAL / ANALYTICAL ISSUES | 12 |
| | 14.1 | Handling of Dropouts or Missing Data | 12 |
| | 14.2 | Pooling of Centers in Multi-Center Studies | 12 |
| | 14.3 | Multiple Comparison / Multiplicity | 12 |
| | 14.4 | Examination of Subgroups. | 12 |
| | 14.5 | Interim Analyses and Data Monitoring. | 13 |
| 15 | REF | ERENCES | 14 |
| 16 | A DD | DENDICES | 1 4 |

| I | JST | OF | In-t | EXT | TA | RI | ES |
|---|-----------|------------|------|-----|----|----|----|
| | / I L J I | <b>\</b> / | | | | | |

# LIST OF APPENDICES


Clovis Oncology 01 March 2021

## ABBREVIATIONS AND SPECIALIST TERMS

AE(s) adverse event(s)

ANC absolute neutrophil count
AST aspartate aminotransferase
ALT alanine aminotransferase

BID twice daily

CEOI concentration at the end of infusion

 $C_{min}$  minimum concentration

CRM cohort review meeting

CR complete response
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

ctDNA circulating cell-free tumor DNA

DLT dose limiting toxicity
ECG electrocardiogram

GCSF granulocyte colony-stimulating factor

IMMU-132 sacituzumab govitecan
MTD maximum tolerated dose

NCI National Cancer Institute

ORR objective response per RECIST

PD progressive disease
PK pharmacokinetic(s)
PR partial response

RP2D Recommended Phase 2 dose

RECIST Response Evaluation Criteria in Solid Tumors

SAE serious adverse event SAP statistical analysis plan

SD stable disease

SI International System of Units

StD standard deviation

TEAE treatment-emergent adverse event

ULN upper limit of normal


## 1 Introduction

This statistical analysis plan (SAP) describes the data summaries and any statistical analyses to be performed to assess the safety, efficacy, and pharmacokinetics (PK) of rucaparib (CO-338) for Clovis Oncology, Inc sponsored clinical study CO-338-098, entitled "SEASTAR: A Phase 1b/2, Open-label, Parallel Arm Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral Rucaparib in Combination with Other Anticancer Agents in Patients with a Solid Tumor." This SAP addresses the Phase 1b portion of Arm B of the study since the study did not continue to Phase 2. Enrollment in Arm B, Phase 1b was halted after 2 dose cohorts, so the analysis plan will be reduced from what was indicated in the protocol in order to support a synoptic clinical study report (CSR). It is anticipated that results for Arm A, which is still ongoing at this time, will be analyzed under a different SAP.

## 2 OVERALL STUDY DESIGN, OBJECTIVES, AND ENDPOINTS

### 2.1 STUDY DESIGN

For the Phase 1b portion of Arm B, the plan estimated 6 to 12 dose-escalation cohorts, with a minimum of 3 patients enrolled in each cohort, followed by an expanded evaluation of the recommended phase 2 dose (RP2D) in up to 10 additional patients. Dose escalation was to follow a 3+3 design.

The initial combination dose consists of oral rucaparib 300 mg twice daily (BID), administered continuously, in combination with IV IMMU-132 6 mg/kg administration on Day 1 and Day 8 of a 21-day cycle. The dose of rucaparib was to be escalated in 100 mg BID increments up to a maximum of 600 mg BID. The dose of IMMU-132 was to be escalated in increments of 2 mg/kg, up to a maximum dose of 10 mg/kg.


Clovis Oncology 01 March 2021

### 2.2 STUDY OBJECTIVES AND ENDPOINTS

Because this study was halted before phase 1b was complete, not all endpoints from the protocol will be analyzed. Table 1 outlines the objectives and endpoints planned per protocol for Phase 1b of Arm B. The final column includes the analyses to be included in the CSR.

Table 1. Primary, Secondary, and Exploratory Objectives and Endpoints for Phase 1b

| Primary Objectives | Primary Endpoints | Included in CSR |
|---|---|---|
| To evaluate the safety and tolerability of rucaparib in combination with IMMU-132 and to determine the maximum tolerated dose (MTD) and/or the RP2D of the combination. | Incidence of AEs, clinical laboratory abnormalities, dose modifications, and listings of ECGs and vital signs | AEs, some clinical<br>laboratories, and<br>dose modifications<br>will be included |
| Secondary Objectives | Secondary Endpoints | |
| To characterize the PK of IMMU-132 and its metabolites when rucaparib and IMMU-132 agent are co-administered. | Plasma concentration at trough (C <sub>min</sub> ) and at the end of infusion (C <sub>EOI</sub> ) | Not included in CSR |
| To evaluate the preliminary efficacy of rucaparib in combination with IMMU-132 in various solid tumors. | Objective response per RECIST v1.1 (ORR) | Included in the CSR |
| <b>Exploratory Objectives</b> | Exploratory Endpoints | |
| To assess tumor tissue biomarkers that correlate with response to the combination. | Not defined in protocol | Not included in CSR |
| To evaluate circulating cell-free tumor DNA (ctDNA) as a molecular marker of response to the combination. | Not defined in protocol | Not included in CSR |
| To evaluate biomarkers associated with resistance to the combination. | Not defined in protocol | Not included in CSR |
| To assess genomic changes over time in plasma and tumor samples. | Not defined in protocol | Not included in CSR |
| To determine steady-state exposure of rucaparib by sparse PK sampling. | Not defined in protocol | Not included in CSR |
| To evaluate the development of anti-drug antibodies (ADAs). | Not defined in protocol | Not included in CSR |


### 2.3 SAMPLE SIZE JUSTIFICATION

For Arm B Phase 1b, it was estimated that up to 55 patients would be enrolled following a standard 3+3 design, dependent upon the occurrence of safety findings, specifically DLTs, observed at the different dose levels. 6 subjects were enrolled before the study was halted.

### 3 GENERAL ANALYSIS CONVENTIONS

Quantitative variables will typically be summarized using frequencies and percentages for appropriate categorizations and may also be summarized using descriptive statistics. For variables summarized with descriptive statistics, the following will be presented: N, mean, standard deviation (StD), median, minimum, and maximum. Categorical variables will be presented using frequencies and percentages.

Baseline is defined as the last measurement on or prior to the first dose of rucaparib administration, unless otherwise specified.

All statistical analyses will be conducted with the SAS® System, Version 9.4 or higher.

#### 3.1 Analysis Populations

The following analysis populations are defined for the study:

**Safety Population**: All patients who have received at least 1 dose of rucaparib or IMMU-132.

**DLT-evaluable Population**: All patients in Phase 1b who have either received at least 80% of the planned doses of rucaparib and both planned infusions of IMMU-132 without having experienced a DLT or who experienced a DLT during Cycle 1. If a patient withdrew from the study without having met any of these criteria, then an additional patient was enrolled in that dose cohort.

**Efficacy Population**: All patients who have received at least 1 dose of rucaparib or IMMU-132 and who have measurable disease per RECIST v1.1 at baseline.

# 4 PATIENT DISPOSITION

Patient disposition will be summarized using frequency counts and the corresponding percentages. The number of patients in each analysis population, number of patients discontinued, and the primary reason for treatment discontinuation will be summarized.


## 5 PROTOCOL DEVIATIONS

Protocol deviations will not be analyzed in Arm B of the SEASTAR study.

## 6 DEMOGRAPHICS AND BASELINE CHARACTERISTICS

All demographic will be summarized for the safety population.

### **6.1 DEMOGRAPHICS**

The demographic variables will be summarized with frequency tabulations and descriptive statistics. The demographic variables presented will include age, height, weight and sex using the following categorizations:

- Age (years):  $\leq 50$ , 51-60, 61-70, 71-80, 81-90, > 90;
- Height (cm):  $\leq 75$ , > 75-100, > 100-125, > 125-150, > 150-175, > 175;
- Weight (kg):  $\leq 50$ , > 50-75, > 75-100, > 100-125, > 125-150, > 150
- Sex: Male, Female

### **6.2** BASELINE CLINICAL CHARACTERISTICS

No baseline disease characteristics will be analyzed in the CSR.

### **6.3** MEDICAL HISTORY

In a change from the protocol, medical history events will not be analyzed.

## 7 DOSE-LIMITING TOXICITIES

A summary of the number of DLTs by dose level and a patient listing of all DLTs will be provided for the patients in the DLT-evaluable population. A DLT is defined at any of the following events occurring in Cycle 1, according to CTCAE version 5.0:

- Grade 3 or greater febrile neutropenia (i.e., fever > 38.3°C with Absolute Neutrophil Count (ANC) < 1.0 × 109/L) of any duration;
- Grade 3 or 4 neutropenia lasting more than 7 days despite granulocyte colonystimulating factor (GCSF) administration; Grade 3 thrombocytopenia (platelets < 50 × 109/L) with significant bleeding or Grade 4 thrombocytopenia (platelets < 25 × 109/L) ≥ 5 days duration;
- Grade 4 anemia (i.e., life-threatening consequences; urgent intervention indicated) or any anemia (regardless of grade or severity) requiring a blood transfusion;
- Any nonhematological  $AE \ge Grade 3$ , with the exception of:


- o Nausea, vomiting, and diarrhea if well controlled by systemic medication and with duration ≤ 48 hrs;
- o Fatigue;
- o Grade 3 alanine aminotransferase (ALT) or aspartate aminotransferase (AST) not accompanied by a concomitant increase in total bilirubin above the upper limit of normal (ULN). Note: any Grade 4 ALT/AST is a DLT.
- Any Grade 3 or greater infusion-related reaction that fails to resolve within 4 hours despite optimal medical management.

## 8 STUDY DRUG EXPOSURE AND COMPLIANCE

The following variables will be summarized:

- Duration of treatment (days)
- Number of dose reductions
- Number of dose interruptions

Duration of treatment will be calculated as 1+ the number of days from earliest study drug start date to date of last study drug discontinuation. Descriptive statistics and frequencies/percentages for appropriate categorizations will be used to summarize study drug exposure variables.

## 9 PRIOR AND CONCOMITANT MEDICATIONS

Prior and concomitant medications will not be analyzed in the CSR.

## 10 EFFICACY ANALYSIS

Efficacy analyses will be performed using the efficacy population.

Overall objective response to treatment according to RECIST v1.1 as assessed by the investigator will be listed along with target lesion measurements and response, non-target lesion response, and assessment of new lesions. Confirmation of a complete response (CR) or partial response (PR) is a response that is maintained and documented on a subsequent tumor assessment no less than 4 weeks after initial response and will be indicated on the listing. Duration of response will also be calculated as the time from the date that a confirmed PR or CR is first recorded until the first date that progressive disease (PD) is documented per RECIST v1.1. Duration of stable disease (SD) will be calculated from the start of treatment to the first PD if the subject had a best response of SD.

A listing of all tumor scan details collected, including ORR, in the clinical database will be provided.


## 11 EXPLORATORY ANALYSIS

No exploratory endpoints will be analyzed in the CSR.

## 12 PHARMACOKINETIC ANALYSIS

PK analyses, including the secondary endpoint, will no longer be included in the CSR due to the early termination of the study.

## 13 SAFETY ANALYSIS

The safety analyses will be performed using the safety population.

### 13.1 ADVERSE EVENTS

Adverse events (AEs) will be classified using the MedDRA classification system. The severity of the toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 whenever possible. Treatment-emergent adverse events (TEAEs) are defined as AEs with onset date on or after the date of first dose of study medication until the date of the last study medication dose plus 28 days. Adverse events will be considered treatment-emergent if all or part of the date of onset of the AE is missing and it cannot be determined if the AE meets the definition for treatment-emergent.

The number and percentage of patients who experienced TEAEs for each system organ class and preferred term will be presented. Multiple instances of the TEAE in each system organ class and multiple occurrences of the same preferred term are counted only once per patient. The number and percentage of patients with at least one TEAE will also be summarized.

The incidence of TEAEs will also be summarized by relationship to study drug according to the following categories: "treatment-related," or "not treatment-related" for each study drug. If a patient experiences multiple occurrences of the same AE with different relationship categories, the patient will be counted once, as a relationship category of treatment-related.

If a patient experiences multiple occurrences of the same AE with different toxicity grades, the patient will be counted once for the maximum (most severe) toxicity grade. AEs with a missing toxicity grade will be presented in the summary table with a toxicity grade of "Missing." For each toxicity grade, the number and percentage of patients with at least one TEAE of the given grade will be summarized.

Separate tables will be presented including but not limited to:

- All TEAEs;
- TEAEs by CTCAE grade;
- Grade 3 or greater TEAEs;


- Treatment-related TEAEs, overall and by categories: CTCAE grade, grade 3 or greater, resulting in dose reduction, resulting in dose interruption, resulting in dose discontinuation, outcome of death;
- Serious TEAEs:
- TEAEs with an outcome of death;
- TEAEs leading to discontinuation of study medication;
- TEAEs resulting in interruption of study medication; and
- TEAEs resulting in reduction, delay, or interruption of study medication.

### 13.2 CLINICAL LABORATORY EVALUATIONS

Clinical laboratory evaluations include the continuous variables for hematology, chemistry, and urinalysis. The laboratory values will generally be presented in International System (SI) units. The on-treatment period will be defined as the time from earliest first dose to 28 days after the last dose of rucaparib or IMMU-132, whichever is last. Hematology values collected will be listed. Descriptive summaries, and all chemistry and urinalysis parameters, mentioned in the protocol will not be included in the analysis.

### 13.3 VITAL SIGNS

Vital signs will not be analyzed in this study.

## 14 STATISTICAL / ANALYTICAL ISSUES

### 14.1 HANDLING OF DROPOUTS OR MISSING DATA

All data will be used to their maximum possible extent, but without any imputations for missing data.

### 14.2 POOLING OF CENTERS IN MULTI-CENTER STUDIES

All centers will be pooled for analysis.

### 14.3 MULTIPLE COMPARISON / MULTIPLICITY

No statistical comparisons will be performed.

### 14.4 EXAMINATION OF SUBGROUPS

Analyses of primary and secondary endpoints may be analyzed by starting dose. No additional subgroup analyses will be performed.


Rucaparib CO-338-098B Statistical Analysis Plan Clovis Oncology 01 March 2021

## 14.5 INTERIM ANALYSES AND DATA MONITORING

No formal interim analyses were planned outside standard Cohort Review Meetings (CRM). CRMs were held for the first 2 dose cohorts and the decision was made to forgo exploration of any other dose cohorts.


Clovis Oncology 01 March 2021

# 15 REFERENCES

1. Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45(2):228-47.


## 16 APPENDICES

### Appendix 1 Response Evaluation Criteria in Solid Tumors

The RECIST guidelines (Version 1.1) are described in Eisenhauer (2009)<sup>1</sup> and at http://www.eortc.be/Recist/Default.htm. A short summary is given below.

#### **Measurable Disease:**

<u>Tumor lesions</u>: measurable lesions are defined as those that can be accurately measured in at least 1 dimension (longest diameter to be recorded) with the following:

- A minimum size of 10 mm by CT scan (CT scan thickness no greater than 5 mm).
- A minimum size of 10 mm caliper measurement by clinical exam (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable).
- A minimum size of 20 mm by chest X-ray.

All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

<u>Malignant lymph nodes</u>: to be considered pathologically enlarged and measurable, a lymph node must be  $\geq 15$  mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be not greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

### Nonmeasurable Disease:

All other lesions (or sites of disease), including small lesions (longest diameter < 10 mm or pathological lymph nodes with  $\ge$  10 to < 15 mm short axis), as well as truly nonmeasurable lesions, are considered nonmeasurable disease. Lesions considered truly nonmeasurable include leptomeningeal disease, ascites, pleural/pericardial effusions, inflammatory breast disease, lymphangitic involvement of skin and lung, and abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.

#### **Bone Lesions**

Bone lesions, cystic lesion, and lesions previously treated with local therapy require particular comment. Bone scan, PET scan, or plain films are not considered adequate imaging techniques to measure bone lesions. However, these techniques can be used to confirm the presence or disappearance of bone lesions.

Lytic bone lesions or mixed lytic—blastic lesions with identifiable soft tissue components that can be evaluated by cross-sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the soft tissue component meets the definition of measurability described above.


Clovis Oncology 01 March 2021

Blastic bone lesions are nonmeasurable.

### **Cystic Lesions**

Lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor nonmeasurable) because they are, by definition, simple cysts.

Cystic lesions thought to represent cystic metastases can be considered as measurable lesions if they meet the definition of measurability described above. However, if noncystic lesions are present in the same patient, these are preferred as target lesions.

### **Lesions with Prior Local Treatment**

Tumor lesions situated in a previous irradiated area or in an area subjected to other locoregional therapy are usually not considered measurable unless there has been demonstrated progression in the lesion.

### **Target Lesions**

All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as target lesions and recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference by which to characterize the objective tumor response.

### **Nontarget Lesions**

RECIST criteria require unequivocal quantification of the changes in tumor size for adequate interpretation of the sum of target lesions. Consequently, when the boundaries of the primary are difficult to delineate, this tumor should not be considered a target lesion.

#### **Guidelines for Evaluation of Measurable Disease**

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination when both methods have been used to assess the antitumor effect of a treatment.


| Evaluation of Target L | Evaluation of Target Lesions |
|---|---|
| Complete Response | Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm. |
| Partial Response | At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. |
| Stable Disease | Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. |
| Progressive Disease | At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. |

Abbreviations: LD = longest diameter; PD = progressive disease.

| <b>Evaluation of Nontarget Lesions</b> | |
|---|---|
| Complete Response | Disappearance of all nontarget lesions and normalization of tumor marker level. |
| Stable Disease/Incomplete<br>Response | Persistence of 1 or more nontarget lesion(s) or/and maintenance of tumor marker level above the normal limits. |
| Progressive Disease | Appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions. |

If tumor markers are initially above the institutional ULN, they must normalize for a patient to be considered a complete responder.

### **Evaluation of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

| <b>Evaluation of Best Overall Response</b> | | | |
|---|---|---|---|
| <b>Target Lesions</b> | Nontarget Lesions | New Lesions | Overall Response |
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |


| Evaluation of Best Overall Response | | | | | |
|---|---|---|---|---|---|
| Target Lesions | | esions | Nontarget Lesions | New Lesions | Overall Response |
| CR | | | Not evaluated | No | PR |
| PR | | | Non-PD or not evaluated | No | PR |
| SD | | | Non-PD or not evaluated | No | SD |
| Not Evaluated | | ıated | Non-PD | No | NE |
| PD | | | Any | Yes or No | PD |
| Any | | | PD | Yes or No | PD |
| Any | | | Any | Yes | PD |
| CR | = | complete response | | | |
| NE | = | not evaluable. | | | |
| PD | = | progressive disease | | | |
| PR | = | partial response | | | |
| SD | = | stable disease | | | |

Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be classified as having symptomatic deterioration. Every effort should be made to document the objective progression, even after discontinuation of treatment.

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When the evaluation of CR depends on this determination, it is recommended that the residual lesion be investigated (fine needle aspiration/biopsy) prior to confirming the complete response status.

### **Confirmatory Measurement/Duration of Response**

### Confirmation

If a complete response (CR) or partial response (PR) is noted, confirmatory scans should be performed at least 4 weeks after response was first documented.

### **Duration of Overall Response**

The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or PD is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started).

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.


Rucaparib CO-338-098B Statistical Analysis Plan Clovis Oncology 01 March 2021

## **Duration of Stable Disease**

Stable disease (SD) is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.
